CLINICAL TRIAL: NCT00721786
Title: Internet Health Research Center: Smoking, Latinos, and the Web
Brief Title: Internet Stop Smoking Study - Phase VI
Acronym: TC4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IWHRC-RFM-SMK-PhVI
Record Dates: First submitted 2008-07-22; First posted 2008-07-24 (Estimated); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Smoking
Keywords: Smoking cessation; Cigarette smoking; Tobacco smoking; Internet interventions; Spanish-speaking
MeSH Terms: conditions — Smoking; Smoking Cessation; Cigarette Smoking; Tobacco Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- San Francisco Internet Stop Smoking Site (Experimental): UCSF/SFGH Internet Stop Smoking Study site
  Internet Stop Smoking site (TC4) with several intervention elements from which the participants may choose as many as they wish
  The links (URLs) to register for the study are:
  English: www.stopsmoking.ucsf.edu Spanish: www.dejardefumar.ucsf.edu
  Interventions: Behavioral: UCSF/SFGH Internet Stop Smoking Study site

INTERVENTIONS:
Behavioral: UCSF/SFGH Internet Stop Smoking Study site — Internet stop smoking site in Spanish and English
  Other Names: The interventions being tested can be accessed online at:; www.stopsmoking.ucsf.edu; www.dejardefumar.ucsf.edu

SUMMARY:
The purpose of this study is to determine the percentage of English- and Spanish-speaking smokers worldwide who can stop smoking using an Internet stop smoking site.

Latinos and non-Latinos are welcome to participate.

We will stop recruitment on March 19, 2011. Participants will be able to use the site until May 19, 2011.

DETAILED DESCRIPTION:
This is Phase VI of a series of clinical trials comparing various Internet methods to help smokers quit via the Internet.

Our previous trials have involved randomized assignment. This trial is a participant preference trial, in which English- and Spanish-speaking smokers will be able to choose the elements of the site which they would like to use to stop smoking.

Smokers who find our link via search engines or listing on other Web sites may choose to enter the study.

Participants must be 18 years old to enter the study. Participants will be followed up at 1, 3, 6, and 12 months after entry into the study to determine whether they have stopped smoking. They will receive an email reminder with a link to our follow-up surveys. We will stop sending these email reminders on May 19, 2011, when the current Website will close.

Participation is totally voluntary. Participants are free not to provide data or to stop participating at any time.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 years old or above)
* must have email
* logging on to our stop smoking Internet site
* providing consent to enter stop smoking study

Exclusion Criteria:

* Younger than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18154 (Actual)
Dates: Start 2008-09; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Smoking abstinence | 1, 3, 6 and 12 month follow-ups
  Not smoking even one cigarette in the past 7 days.

SECONDARY OUTCOMES:
Depression | 1, 3, 6, and 12 month follow-ups
  Center for Epidemiological Studies Depression scale

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo F. Muñoz, Ph.D., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco SFGH Psychiatry, San Francisco, California, United States

REFERENCES:
- [Background] Munoz RF, Barrera AZ, Delucchi K, Penilla C, Torres LD, Perez-Stable EJ. International Spanish/English Internet smoking cessation trial yields 20% abstinence rates at 1 year. Nicotine Tob Res. 2009 Sep;11(9):1025-34. doi: 10.1093/ntr/ntp090. Epub 2009 Jul 29. PMID 19640833
- [Background] Munoz RF, Lenert LL, Delucchi K, Stoddard J, Perez JE, Penilla C, Perez-Stable EJ. Toward evidence-based Internet interventions: A Spanish/English Web site for international smoking cessation trials. Nicotine Tob Res. 2006 Feb;8(1):77-87. doi: 10.1080/14622200500431940. PMID 16497602
- [Background] Torres LD, Barrera AZ, Delucchi K, Penilla C, Perez-Stable EJ, Munoz RF. Quitting smoking does not increase the risk of major depressive episodes among users of Internet smoking cessation interventions. Psychol Med. 2010 Mar;40(3):441-9. doi: 10.1017/S0033291709990560. Epub 2009 Jul 23. PMID 19627638
- [Background] Barrera AZ, Perez-Stable EJ, Delucchi KL, Munoz RF. Global reach of an Internet smoking cessation intervention among Spanish- and English-speaking smokers from 157 countries. Int J Environ Res Public Health. 2009 Mar;6(3):927-40. doi: 10.3390/ijerph6030927. Epub 2009 Feb 26. PMID 19440423
- [Derived] Munoz RF, Aguilera A, Schueller SM, Leykin Y, Perez-Stable EJ. From online randomized controlled trials to participant preference studies: morphing the San Francisco Stop Smoking site into a worldwide smoking cessation resource. J Med Internet Res. 2012 Jun 27;14(3):e64. doi: 10.2196/jmir.1852. PMID 22739225
- [Derived] Leykin Y, Aguilera A, Torres LD, Perez-Stable EJ, Munoz RF. Interpreting the outcomes of automated internet-based randomized trials: example of an International Smoking Cessation Study. J Med Internet Res. 2012 Feb 7;14(1):e5. doi: 10.2196/jmir.1829. PMID 22314016